CLINICAL TRIAL: NCT03971773
Title: PSYCHOLOGICAL CARE AND HYPNOSIS IN PATIENTS WITH CANCER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-A00472-53; 2018-A00472-53 (Other: Assistance Publique Hôpitaux de Marseille)
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Hypnosis and Cancer
MeSH Terms: conditions — Neoplasms | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient ongoing hypnosis sessions (Experimental)
  Interventions: Other: hypnosis

INTERVENTIONS:
Other: hypnosis — patient with cancer will undergo sessions of hypnosis

SUMMARY:
The general aim of the research that we propose to implement is to study the potential benefits of hypnosis in the psycho-social care of patients with cancer. The main goal of this study is to measure the effects of hypnosis sessions on quality of life, anxiety and patient adjustment strategies. The effects of these interventions will be the subject of quantitative measurement via standardized scales in pre- and post-intervention situations of the potential effects of hypno-therapeutic intervention in cancer patients and

ELIGIBILITY:
Inclusion Criteria:

* Patient with any kind of cancer and followed by a psychologist

Exclusion Criteria:

* Patient with neurological trouble
* Patient with psychiatric decompassation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2021-04-18 (Estimated); Study Completion 2022-04-18 (Estimated)

PRIMARY OUTCOMES:
quality of life scale | 36 months
  QLQC30 assessment

SECONDARY OUTCOMES:
anxiety scales | 36 months
  Edmonton Symptom Assessment System

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance publique hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided